CLINICAL TRIAL: NCT04650698
Title: The Effect of Tranexamic Acid on Calculated Total Blood Loss in Patients Undergoing Revision Shoulder Arthroplasty
Brief Title: TXA in Revision Total Shoulder Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment rate was slower than anticipated.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-01617
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Arthropathy Shoulder
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Neither the anesthesiologist or surgeon will be blinded to the patient's group assignment, as they will be the one performing the treatment. All other stakeholders (patient, other caregivers, and research staff collecting the data) will be blinded to the patient's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (TXA) Injection (Experimental): Participants scheduled for Revision Total Shoulder Arthroplasty (TSA) will receive two injections of TXA.
  Interventions: Drug: Tranexamic acid (TXA) injection
- Control - No Tranexamic acid (TXA) Injection (No Intervention): Participants scheduled for Revision Total Shoulder Arthroplasty (TSA) won't receive any injections TXA.

INTERVENTIONS:
Drug: Tranexamic acid (TXA) injection — IV, Total Dosage: 2 grams (1 gram before surgical incision + 1 gram, 3 hours after first dose)
  Other Names: TXA
  Arms: Tranexamic acid (TXA) Injection

SUMMARY:
This is a phase IV, randomized, single-blind, single-center study comparing calculated total blood loss, surgical drain output and hematoma formation in patients who receive 2 doses of Tranexamic Acid (TXA) versus control group undergoing revision total shoulder arthroplasty. Patients will be randomized to either receive 2 doses of IV TXA, first dose prior to surgical incision and second dose given 3 hours later or to the control group, where no TXA will be administered.

DETAILED DESCRIPTION:
The objectives of the study are to compare the effectiveness of IV TXA on reducing calculated total blood loss, surgical drain output and hematoma formation in patients undergoing revision total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old
2. Patients younger than 90 years old
3. Patients undergoing scheduled revision total shoulder arthroplasty
4. Patients who consent to be randomized

Exclusion Criteria:

1. Patients younger than 18
2. Patients older than 90 years old
3. Patients who are pregnant or breast-feeding women
4. Patients who are allergic to tranexamic acid
5. Patients with proximal humerus fracture or fracture sequelae
6. Patients who use estrogen containing medications (i.e. oral contraceptive pills)
7. Patients who have acquired disturbances of color vision
8. Patients with a history of any of the following diagnosis: '

   * Subarachnoid hemorrhage
   * Active intravascular clotting
   * Severe pulmonary disease (FEV <50% normal)
   * Plasma creatinine > 115 μmol/L in males, > 100 μmol/L in females, or hepatic failure)
   * (Renal impairment serum creatinine > 1.5 times the upper limit of normal NYU)
   * Preoperative anemia [Hemoglobin (Hb) < 11g/dL in females, Hb < 12 g/dL in males]
9. Patients who refuse blood products
10. Patients undergoing hormone replacement therapy
11. Patients with diagnosed or self-reported cognitive dysfunction;
12. Patients who are unable to understand or follow instructions;
13. Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
14. Patients with BMI over 50
15. Any patient that the investigators feel cannot comply with all study related procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hertling, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Orthopedic Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Uchenna.Umeh@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Started | 12 | 7
Completed | 10 | 5
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (6.685) | 62 (8.98) | 63 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 2 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Calculated Total Blood Loss
Description: The volume of perioperative blood loss will be determined on the basis of the blood volume and change in hemoglobin from preoperatively to 1 day postoperatively. The volume of total perioperative blood loss will be determined according to the following formula:
  Total blood loss (ml) = 1000 x 〖Hb〗_loss/〖Hb〗_i
Time Frame: up to 24 hours post-op
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Number analyzed (Participants) | 10 | 5
Milliliters | 0.5952 (0.3312) | 0.8306 (0.3641)

2. Primary Outcome: Total Surgical Drain Output
Description: The floor nurse will also document the amount of blood in the indwelling hemovac surgical drain placed in the operative shoulder joint up to 24 hours. The total surgical drain output will be calculated after 24 hours.
Time Frame: up to 24 hours post-op
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Number analyzed (Participants) | 10 | 5
Milliliters | 101.5 (88.43) | 153 (129)

3. Secondary Outcome: Number of Participants With Presence of Hematoma
Description: Surgeon will assess for presence of hematoma at the 2-week follow up visit.
Time Frame: 2 weeks post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Number analyzed (Participants) | 10 | 5
Participants | 1 | 0

4. Secondary Outcome: Number of Participants Who Needed a Post-op Blood Transfusion
Time Frame: 2 weeks post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Number analyzed (Participants) | 10 | 5
Participants | 0 | 0

5. Secondary Outcome: Average Operative Time
Time Frame: During operation, up to 4 hours
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
Number analyzed (Participants) | 10 | 5
minutes | 104.6 (26.12) | 130.4 (37.58)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Tranexamic Acid (TXA) Injection | Control - No Tranexamic Acid (TXA) Injection
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04650698/Prot_SAP_000.pdf